CLINICAL TRIAL: NCT04427787
Title: A Phase II Trial Aiming to Assess the Safety and Activity of the Combination of Cabozantinib Plus Lanreotide in Gastroenteropancreatic (GEP) and Thoracic Neuroendocrine Tumor (NET): The LOLA Trial
Brief Title: A Trial Aiming to Assess the Safety and Activity of the Combination of Cabozantinib Plus Lanreotide in GEP and NET
Acronym: LOLA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-004506-10
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Well Differentiated Neuroendocrine Neoplasm; Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — cabozantinib; lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib+lanreotide (Experimental): Cabozantinib will be administered orally at a dose of 60 mg/day continuously in combination with Lanreotide 120 mg injection every 28 days. Both treatments will start the same day
  Interventions: Drug: Cabozantinib; Drug: Lanreotide

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib will be administered orally at a dose of 60 mg/day
  Other Names: Cabometyx
Drug: Lanreotide — Lanreotide will be administrated 120 mg injection every 28 days
  Other Names: IPSTYL

SUMMARY:
A Phase II trial aiming to assess the safety and activity of the combination of cabozantinib plus lanreotide in gastroenteropancreatic (GEP) and thoracic neuroendocrine tumor (NET): The LOLA trial

DETAILED DESCRIPTION:
Phase II, multicenter, open-label, non-comparative, non-randomized study with three-stage design

ELIGIBILITY:
Inclusion Criteria:

* voluntary written informed consent obtained before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care;
* Patients with unresectable, advanced or metastatic neuroendocrine well differentiated GEP-NET (pancreatic NET (G2-G3), Small Intestinal NET, stomach NET, rectum NET) with Ki67 10%.
* Patients with unresectable, advanced or metastatic neuroendocrine well differentiated thoracic NET (typical and atypical lung NET, thymus NET)
* Patients with unresectable, advanced or metastatic neuroendocrine well differentiated unknown primary NET with Ki67 10%.
* Locally advanced or metastatic disease documented as progressive by RECIST v1.1. on CT-scan or MRI at baseline and within 12 months prior to baseline.
* disease that is not amenable to surgery with curative intent;
* presence of at least one measurable target lesion for further evaluation according to RECIST v1.1;
* age ≥18 years;
* eastern Cooperative Oncology Group (ECOG) performance status 0 or 1(see APPENDIX I)
* Octreoscan and/or positron emission tomography (PET) 68 Gallium-Dotatoc (68Ga) positive and/or Immuno-histochemistry (IHC) for SSTR2;
* advanced GEP, thoracic and unknown origin NET limited to treatment naïve patients or who have received maximum 1 prior systemic regimen for metastatic disease (biological therapy, chemotherapy or somatostatin analogs, including PRRT);
* Prior PRRT therapy must be completed at least 6 months prior to enrollment;
* Prior treatment with somatostatin analogs, biologic therapy, immunotherapy, chemotherapy, investigational agent for malignancy, and/or radiation must be completed at least 28 days prior to registration;
* Prior treatment with hepatic artery embolization (including bland embolization, chemoembolization, and selective internal radiation therapy) or ablative therapies must be completed at least 28 days prior to registration;
* Prior treatment with cabozantinib or lanreotide are not allowed;
* Patients should have resolution of any toxic effects of prior therapy (except alopecia and fatigue) to National Cancer Institute (NCI) CTCAE, version 5.0, grade 1 or less
* Patients must have completed any major surgery at least two months prior to registration and any minor surgery (including uncomplicated tooth extractions) at least 28 days prior to registration; complete wound healing from major surgery must have occurred at least 1 month prior to registration, and complete wound healing from minor surgery must have occurred at least 7 days prior to registration
* Non-functioning tumors;
* all of the following laboratory test findings:
* Hemoglobin > 9 g/dL (5.6 mmol/L)
* White blood cell count (WBC) > 2,000/mm3
* Neutrophils > 1,500/mm3
* Platelets > 100,000/mm3
* liver enzymes (AST or ALT)< 3 x ULN (< 5 x ULN if liver metastases are present)
* Total Bilirubin < 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Adequate renal function, based upon meeting the following laboratory criteria:

  1. Serum creatinine ≤ 1.5 ´ upper limit of normal (ULN) or calculated creatinine clearance ≥ 40 mL/min using the Cockcroft-Gault equation: (140 - age) × weight (kg)/(serum creatinine × 72 [mg/dL]) for males. (For females multiplied by 0.85)
  2. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.1 mg/mmol) or 24-hour urine protein < 1 g
* Lipase < 2.0 x the upper limit of normal and no radiologic or clinical evidence of pancreatitis
* prothrombin time - international normalized ratio/ partial thromboplastin time (PT/PTT) ≤ 1.5 x upper limit of normal.
* Availability of a representative formalin-fixed paraffin-embedded fractional Fokker-Planck equation (FFPE) tumor specimen collected before starting treatment with cabozantinib and lanreotide that enables the definitive diagnosis of NET (the archival specimen must contain adequate viable tumor tissue to enable candidate biomarkers status; the specimen may consist of a tissue block or at least 10 unstained serial sections with 3 microns of thickness; for core needle biopsy specimens, at least two cores should be available for evaluation)
* Female subjects of childbearing potential must not be pregnant at screening
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception with a failure rate of < 1% per year (eg, barrier methods, including male condom or female condom with spermicidal gel, intrauterine devices, surgical male or female sterilisation) during the study and for 4 months after the last dose of study treatment
* Female subject is either: post-menopausal for at least one year before the screening visit, or surgically sterilized, or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject, even if surgically sterilized (ie, status postvasectomy), agrees to use an acceptable method for contraception during the entire study treatment period through 4 months after the last dose of cabozantinib.
* Patients must be accessible for treatment and follow up as well as they must be willing and capable to comply with the requirements of the study

Exclusion Criteria:

* Patients with undifferentiated, poorly differentiated GEP-NET, Thoracic or unknown primary NET;
* Previous therapy for advanced disease > 1 line; any medical adjuvant treatment must have been stopped at least six months before entry into the study;
* Prior treatment with dose superior or equal to 120 mg per month of lanreotide;
* Prior treatment with cabozantinib;
* Prior treatment with any other tyrosine kinase inhibitors or anti-VEGF angiogenic inhibitors is permitted. Prior treatment with non-VEGF-targeted angiogenic inhibitors such as Everolimus is permitted;
* Patients who stopped Everolimus or tyrosine kinase inhibitors or anti-VEGF angiogenic inhibitors treatment less than 4 weeks prior to the start of the study;
* Patients with concomitant treatment with Interferon;
* Patients previously treated with chemotherapy, loco-regional therapy (e.g., chemoembolization) or interferon with last administration less than 4 weeks prior to the start of the study or with toxicity not resolved to less or equal grade 1 at the start of the study;
* PRRT therapy with last administration less than 6 months prior to inclusion in the study or with toxicity not resolved to less or equal grade 1 at the start of the study;
* diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri;
* history of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA see Appendix II);
* prolongation of QT interval: Cabozantinib should be used with caution in patients with a history of QT interval prolongation, patients who are taking antiarrhythmics, or patients with relevant pre-existing cardiac disease, bradycardia, or electrolyte disturbances (e.g., hypokaliemia, family history of long QT Syndrome). Corrected QT interval calculated by the Fridericia formula (QTcF) 500 ms within 28 days before registration should be shown. Only subjects with a baseline QTcF 500 ms are eligible for the study.

Note: If the QTcF was > 500 ms in the first ECG, a total of 3 ECGs were to be performed. If the average of these 3 consecutive results for QTcF was ≤ 500 ms, the subject met eligibility in this regard.

* history of aneurysms and arterial dissections. The use of VEGF pathway inhibitors in patients with or without hypertension may favor the formation of aneurysms and / or arterial dissections. Before starting cabozantinib, this risk must be carefully considered in patients with risk factors such as hypertension or history of aneurysm.
* poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90 millimeters of mercury(mmHg)];
* history of cerebrovascular accidents, including transient ischemic attack (TIA), history of thromboembolic events (including pulmonary embolism) or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible;
* concomitant anticoagulation at therapeutic doses with oral anticoagulant (eg. Warfarin, direct thrombin and factor 10a inhibitors) or platelet inhibitors (eg. clopidogrel);
* major surgery or trauma within 28 days prior to study entry; the presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement are not considered to be major surgery);
* known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before the start of the study. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of inclusion;
* With the exclusion of inhaled steroids, chronic treatment with corticosteroids with dose superior of 10 mg/day methylprednisolone equivalent must be avoided;
* evidence of active bleeding or bleeding diathesis and/or clinically-significant GI bleeding within 6 months before the first dose of study treatment; 3 months for pulmonary hemorrhage and patients with tumor invading or encasing any major blood vessels;
* patients with GI disorders associated with a high risk of perforation or fistula formation;
* major surgery within 2 months before to registration. Complete healing from major surgery must have occurred 1 month before registration. Complete healing from minor surgery (eg, simple excision, tooth extraction) must have occurred at least 7 days before registration. Subjects with clinically relevant complications from prior surgery are not eligible
* subjects with clinically relevant ongoing complications from prior radiation therapy
* positive test for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness;
* patients with complicated, symptomatic untreated lithiasis of the bile ducts;
* any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, provision of informed consent, or compliance to study procedures;
* previous or ongoing treatment (except for adjuvant therapies) with any of the following anti-cancer therapies: chemotherapy, immunotherapy, target therapies, investigational therapy or hormonal therapy within 28 days or five half-lives of a drug (whichever is longer) prior to the first dose of cabozantinib plus lanreotide;
* inability to swallow tablets;
* rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* previously identified allergy or hypersensitivity to to the study drugs and/or their excipients of the study treatment formulations;
* concomitant use of strong inhibitor of CYP3A4 (i.e. information reported in session 4.5 of the protocol)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 42 months
  according to RECIST, v1.1 defined as complete response or partial response after treatment administration
Primary Safety Endpoint | 42 months
  Adverse Events (AE) grade 3-5 according to NCI-CTCAE v5.0 grade

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 42 months
  defined as the time from first day of treatment administration until progression disease according to RECIST v 1.1 or death for every cause, whichever occurred first.
Safety Endpoint | 42 months
  Adverse Event (AE) all grade according to NCI-CTCAE v5.0 grade
Clinical effectiveness endpoint | 42 months
  Overall Survival (OS) defined as the time from first treatment administration until death whichever cause
Exploratory objectives analysis | 42 months
  the investigation of immunohistochemical tissue expression level of Mesenchymal Epithelial Transition (MET), AXL, vascular endothelial growth factor (VEGFR2) proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pusceddu, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Result] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Blumberg J, Ruszniewski P; CLARINET Investigators. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Jul 17;371(3):224-33. doi: 10.1056/NEJMoa1316158. PMID 25014687
- [Result] Susini C, Buscail L. Rationale for the use of somatostatin analogs as antitumor agents. Ann Oncol. 2006 Dec;17(12):1733-42. doi: 10.1093/annonc/mdl105. Epub 2006 Jun 26. PMID 16801334
- [Result] Krantic S, Goddard I, Saveanu A, Giannetti N, Fombonne J, Cardoso A, Jaquet P, Enjalbert A. Novel modalities of somatostatin actions. Eur J Endocrinol. 2004 Dec;151(6):643-55. doi: 10.1530/eje.0.1510643. PMID 15588232
- [Result] Chalabi M, Duluc C, Caron P, Vezzosi D, Guillermet-Guibert J, Pyronnet S, Bousquet C. Somatostatin analogs: does pharmacology impact antitumor efficacy? Trends Endocrinol Metab. 2014 Mar;25(3):115-27. doi: 10.1016/j.tem.2013.11.003. Epub 2014 Jan 7. PMID 24405892
- [Result] Rai U, Thrimawithana TR, Valery C, Young SA. Therapeutic uses of somatostatin and its analogues: Current view and potential applications. Pharmacol Ther. 2015 Aug;152:98-110. doi: 10.1016/j.pharmthera.2015.05.007. Epub 2015 May 5. PMID 25956467
- [Result] Pola S, Cattaneo MG, Vicentini LM. Anti-migratory and anti-invasive effect of somatostatin in human neuroblastoma cells: involvement of Rac and MAP kinase activity. J Biol Chem. 2003 Oct 17;278(42):40601-6. doi: 10.1074/jbc.M306510200. Epub 2003 Aug 5. PMID 12902325
- [Result] Azar R, Najib S, Lahlou H, Susini C, Pyronnet S. Phosphatidylinositol 3-kinase-dependent transcriptional silencing of the translational repressor 4E-BP1. Cell Mol Life Sci. 2008 Oct;65(19):3110-7. doi: 10.1007/s00018-008-8418-2. PMID 18810319
- [Result] Raymond E, Dahan L, Raoul JL, Bang YJ, Borbath I, Lombard-Bohas C, Valle J, Metrakos P, Smith D, Vinik A, Chen JS, Horsch D, Hammel P, Wiedenmann B, Van Cutsem E, Patyna S, Lu DR, Blanckmeister C, Chao R, Ruszniewski P. Sunitinib malate for the treatment of pancreatic neuroendocrine tumors. N Engl J Med. 2011 Feb 10;364(6):501-13. doi: 10.1056/NEJMoa1003825. PMID 21306237
- [Derived] Corti F, Brizzi MP, Amoroso V, Giuffrida D, Panzuto F, Campana D, Prinzi N, Milione M, Cascella T, Spreafico C, Randon G, Oldani S, Leporati R, Scotto G, Pulice I, Stocchetti BL, Porcu L, Coppa J, Di Bartolomeo M, de Braud F, Pusceddu S. Assessing the safety and activity of cabozantinib combined with lanreotide in gastroenteropancreatic and thoracic neuroendocrine tumors: rationale and protocol of the phase II LOLA trial. BMC Cancer. 2023 Sep 26;23(1):908. doi: 10.1186/s12885-023-11287-2. PMID 37752423